CLINICAL TRIAL: NCT06645860
Title: Silver Modified Atraumatic Restorative Technique (SMART) With Different Modifications in Asymptomatic Deep Carious Lesions of Primary Molars.
Brief Title: SMART With Different Modifications in Asymptomatic Deep Carious Lesions of Primary Molars.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Hilal Ozturk, Research Assistant, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanakkaleOMU5616
Record Dates: First submitted 2024-04-05; First posted 2024-10-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Caries; Dentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver Diamine Fluoride+Potassium Iodide+Led Light (Experimental): Following the silver diamine fluoride and potassium iodide application, LED light will be applied for 20 seconds.
  Interventions: Procedure: SDF+KI+LED Light 20s; Procedure: SDF+KI
- Silver Diamine Fluoride(Control) (Other): Only silver diamine fluoride and potassium iodide solution will be applied.
  Interventions: Procedure: SDF+KI

INTERVENTIONS:
Procedure: SDF+KI+LED Light 20s — After the silver diamine fluoride (SDF) and potassiım iodide (KI) application, 20-second LED light will be applied to the cavity.
  Arms: Silver Diamine Fluoride+Potassium Iodide+Led Light
Procedure: SDF+KI — Silver diamine fluoride (SDF) and potassium iodide(KI) will be applied.

SUMMARY:
This study aimed to evaluate the clinical success of the 'Silver Modified Atraumatic Restorative Technique '(SMART) with different modifications in asymptomatic deep carious lesions of primary molars.

DETAILED DESCRIPTION:
The SMART technique, which stands for "Silver Modified Atraumatic Restorative Treatment," combines the use of Silver Diamine Fluoride (SDF) with atraumatic restorative treatment methods to manage dental caries.SDF helps strengthen the tooth structure and arrests caries, while atraumatic restorative treatment utilizes high-viscosity glass ionomer cements to remove decayed tissue and repair the tooth with minimal invasion.

Patients between the ages of 4-9 who meet ICDAS II (International Caries Detection and Assessment System) 4-5-6 criteria and need restoration of asymptomatic primary molars with unilateral or multifaceted carious cavities will be included. Volunteers will be randomly divided into 2 groups and the treatments of primary molars will be completed using SMART, SMART + LED light techniques.The teeth in all groups will be cleaned of decay using an excavator first, and then Diagnodent values will be checked.

Group 1 (SMART only): 1 drop of SDF solution will be applied to the cavity for 1 minute with a rubbing motion using a bond brush. Then potassium iodide solution will be applied to prevent discoloration. Following the application, the lesion will be washed with water for 10 seconds and the unreacted SDF solution will be removed from the cavity with cotton pellets, leaving a moist shiny surface.

Group 2: (SMART + LED): 1 drop of SDF will be applied to the cavity for 1 min by rubbing the solution. Then LED light (D-Light Pro, GC Europe) will be applied for 20 s in continuous mode from a distance of approximately 1 cm. The following procedure will be the same as SMART only group.

Following SDF applications and activation, 2 weeks later all groups will be checked by diagnodent and restored with high viscosity glass ionomer cements (EQUIA Forte HT, GC, Tokyo, Japan) in accordance with the manufacturers instructions, and the restoration will be covered with a sealing agent (EQUIA Forte Coat, GC, Tokyo, Japan).

Before the procedure, demographic and dental data of the child volunteer, such as age, gender, brushing frequency, and number of teeth treated, will be recorded.

The US Public Health Service criteria (retention,anatomical form, surface roughness, , secondary caries, marginal discoloration and marginal integrity) and Modified FDI criteria will be used for clinical evaluation of restorations. The restorations will be evaluated clinically and radiologically at baseline 3., 6. and 12. months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and parents of the patients who accept to participate and sign the informed consent.
2. Children between the ages of 4-9
3. Healthy children without a history of serious systemic conditions necessitating chronic use of medications.
4. Children whose dental examination reveals at least one untreated asymptomatic cavitated carious lesion (ICDAS II index: code 4,5,6) affecting primary molars.
5. Absence of former history of spontaneous pain from the offending tooth/teeth.
6. Patients with an appropriate level of cooperation to complete treatment under clinical conditions.
7. Teeth are in a restorable condition.
8. Natural exfoliation of primary teeth to be treated should not be expected within two years.

Exclusion Criteria:

1. Patients and parents of the patients who does not accept to participate and sign the informed consent
2. Patients with proven allergy to silver compounds or any component of dental materials to be applied.
3. Patients with special health care needs or any medical conditions.
4. Primary molar teeth with excessive crown damage that cannot be restored.
5. Primary molar teeth in which bone loss exceeds 1/3 of the roots.
6. Primary molar teeth that have previously undergone root canal treatment or pulpotomy treatment.
7. Presence of internal/external and root resorption in primary teeth to be treated.
8. Root fracture, ankylosis or mobility in the primary teeth to be treated.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
1.Change from 3 months to 12 months regarding "Anatomic form" | 3-month,6-month,12 month
  alpha: The general contour of the restorations follows the contour bravo: the general contour of the restoration does not follow the contour of the tooth charlie: The restoration has an overhang does
Change from 3 months to 12 months regarding "Marginal adaptation" | 3-month,6-month,12 month
  alpha: Explorer does not catch or has one-way catch when drawn across the restoration/tooth interface bravo: explorer falls into crevice drawn across the restoration/tooth interface charlie: Dentin or base is exposed along the margin
Change from 3 months to 12 months regarding "Surface roughness" | 3-month,6-month,12 month
  alpha: the surface of the restoration does not have any surface defects bravo: the surface of the restoration has minimal surface defects charlie: the surface of the restoration has severe surface defects
Change from 3 months to 12 months regarding "Marginal staining" | 3-month,6-month,12 month
  alpha: there is no discoloration between the restorations and tooth bravo: there is discoloration on less than half of the circumferential margin charlie: there is discoloration on more than half of the circumferential margin
Change from 3 months to 12 months regarding "Retention" | 3-month,6-month,12 month
  alpha: intact bravo: chipped/loss of material charlie: complete loss of crown
Change from 3 months to 12 months regarding "Incisal wear" | 3-month,6-month,12 month
  alpha: intact bravo: wear of occlusal surface without tooth surface exposure charlie: wear of occlusal surface with tooth surface exposure
Functional properties according to revised FDI (World Dental Federation) criteria. | 3-month,6-month,12 month
  Functional properties:
  F2: Marginal adaptation measured by visual examination, short air drying, 250 μm probe.
  F3:Proximal contact point measured by visual examination and 25/50/100 μm blades.
  F4: Form and contour measured by visual examination. F5: Occlusion and occlusal wear measured by visual examination and articulation paper.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Biological properties according to revised FDI criteria. | 3-month,6-month,12 month
  Biological properties:
  B1: Caries at restoration margin (CAR) measured by visual examination, short air drying, and 250 μm probe.
  B2: Dental hard tissue defects at restoration margin measured by visual examination.
  B3: Postoperative hypersensitivity reported by patient and pulp status tested with cold stimulus.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Aesthetic properties according to revised FDI criteria. | 3-month,6-month,12 month
  Aesthetic properties:
  A1: Surface luster and surface texture measured by visual examination and short air drying.
  A2: Marginal staining measured by visual examination and short air drying. A3: color match measured by visual examination. Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Kepez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In this study, we are committed to sharing our findings while ensuring the privacy and confidentiality of our participants. Therefore, we will only be disseminating aggregated statistical results derived from the data, rather than individual participant data.